CLINICAL TRIAL: NCT06650748
Title: Multigene Risk Score Combined With Ki-67 Dynamic Assessment in Stratified Neoadjuvant Endocrine Therapy Treatment With or Without CDK4/6 Inhibitors in HR+/HER2- Breast Cancer: a Randomize-controlled Study
Brief Title: Multigene Risk Score Combined With Ki-67 Dynamic Assessment in Stratified Neoadjuvant Endocrine Therapy Treatment With or Without CDK4/6 Inhibitors in HR+/HER2- Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Tao OUYANG, Professor, Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OBU-BC-II-164
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer; Early-stage Breast Cancer
Keywords: Early-stage Breast Cancer; neoadjuvant endocrine therapy; CDK4/6; HR+/HER2-
MeSH Terms: conditions — Breast Neoplasms | interventions — dalpiciclib; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1 (Experimental): gene high-risk according to Epclin who are insensitive to single-agent AI treatment for two weeks
  Interventions: Drug: Dalpiciclib; Drug: Letrozole
- Arm 2 (Experimental): gene high-risk according to Epclin who are sensitive to single-agent AI treatment for two weeks and gene low-risk according to Epclin who are insensitive to single-agent AI treatment for two weeks, randomly assigned to letrozole treatment arm
  Interventions: Drug: Letrozole
- Arm 3 (Experimental): gene high-risk according to Epclin who are sensitive to single-agent AI treatment for two weeks and gene low-risk according to Epclin who are insensitive to single-agent AI treatment for two weeks, randomly assigned to Dalpiciclib and letrozole treatment arm
  Interventions: Drug: Dalpiciclib; Drug: Letrozole
- Arm 4 (Experimental): gene low-risk according to Epclin who are sensitive to single-agent AI treatment for two weeks
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Dalpiciclib — Dalpiciclib, oral administration, 125g each time, once daily, days 1-21, with a 28-day cycle (3 weeks on/1 week off). Continuous medication for 6 cycles, or disease progression, intolerable toxicity, withdrawal from the study for any reason or death, whichever occurs first; or after researcher's judgement, patient would no longer benefit from the treatment.
  Arms: Arm 1; Arm 3
Drug: Letrozole — 2.5 mg, oral, once daily (continuously), with a 28-day cycle. Continuous medication for 6 cycles, or disease progression, intolerable toxicity, withdrawal from the study for any reason or death, whichever occurs first. Refer to drug instructions for specific usage

SUMMARY:
This is a prospective, single-center, randomize-controlled study. The purpose of this study is to evaluate the efficacy of neoadjuvant CDK4/6 inhibitors in patients with high-risk EPclin multigene risk analysis and non-response to Ki-67 2W, and to explore predictive biomarkers for sensitivity to CDK4/6 inhibitor therapy.

DETAILED DESCRIPTION:
China is a country with a high incidence of breast cancer. For operable hormone receptor-positive (HR+) / human epidermal growth factor receptor 2-negative (HER2-) breast cancer, traditional neoadjuvant chemotherapy often fails to achieve clinical complete response (CCR) and has poor tolerability. Endocrine therapy plays a significant role in the treatment of advanced and early-stage HR+/HER2- breast cancer, but its efficacy in neoadjuvant settings needs further exploration. Studies have shown that the CCR and breast conservation rate of neoadjuvant endocrine therapy for HR+/HER2- breast cancer are similar to those of neoadjuvant chemotherapy, with lower toxicity. Therefore, by precisely stratifying the recurrence risk of HR+/HER2- patients and treating them according to different risk levels, the response rate to neoadjuvant endocrine therapy can be further improved, which would be more beneficial for the patients. With the clinical application of CDK4/6 inhibitors, the effectiveness of neoadjuvant endocrine therapy is expected to be enhanced.

In PALLET study, the combination of palbociclib and letrozole significantly inhibited Ki-67 expression, leading to a higher number of patients achieving a state of cell cycle arrest (CCCA) (defined as Ki-67≤2.7%). NeoMONARCH study suggests that a regimen containing abemaciclib is significantly superior to anastrozole monotherapy, with statistical significance (P < 0.001). The NeoPAL and CORALLEEN studies indicate that neoadjuvant endocrine therapy with palbociclib or ribociclib is comparable in efficacy to neoadjuvant chemotherapy, yet has fewer side effects.

EndoPredict (12-gene assay, EPclin) is a second-generation multigene testing scoring tool that combines the molecular biological status of the tumor with clinical factors (tumor size and lymph node status). For early-stage HR+/HER2- breast cancer patients, the EPclin test result helps to distinguish between low and high recurrence risk populations, allowing for a more precise assessment of patient prognosis. In the validation study for premenopausal patients, a total of 385 patients with stage ≤pT3 and pN0~1, who received only endocrine therapy for ER+/HER2- early invasive breast cancer, were enrolled. The results showed that the 10-year distant recurrence-free survival (DRFS) rate for patients in the EPclin low-risk group reached 97%, while the 10-year DRFS rate for the EPclin high-risk group was 76% (P=0.004). For postmenopausal patients, the prognostic value of EPclin was independently validated through the ABCSG6&8 study. The study included 1,702 patients with ER+/HER2- early invasive breast cancer who underwent surgery and received only five years of endocrine therapy. The results showed that the 10-year distant recurrence rate for patients in the EPclin low-risk group was 4%, while the 10-year distant recurrence rates for patients in the EPclin high-risk group were 28% and 22% (P<0.001). A retrospective analysis of ABCSG-34 demonstrated that for patients undergoing neoadjuvant endocrine therapy, the application of EPclin for prognostic assessment revealed a negative correlation between risk levels and residual cancer burden (RCB). That is, among patients receiving neoadjuvant endocrine therapy (NET), a higher proportion of low-risk patients compared to high-risk patients ultimately had an RCB of 0-I.

This study focuses on early-stage HR+/HER2- breast cancer, conducting recurrence risk analysis through EPclin multigene testing, and integrating the dynamic changes of Ki67 after two weeks of neoadjuvant endocrine therapy. Patients are risk-stratified and treated with or without CDK4/6 inhibitors. The study explores the improvement in PEPI scores after surgery and analyzes the effectiveness of multigene testing combined with Ki67 dynamic changes as a predictor for the efficacy of CDK4/6 inhibitor treatment in HR+/HER2- breast cancer with high recurrence risk and insensitivity to endocrine therapy. The study also seeks to explore methods for predicting sensitivity to CDK4/6 inhibitor treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Females aged 18 to 70 years;
2. Patients with histologically confirmed HR+/HER2- invasive breast cancer that is sensitive to endocrine therapy. Tumor diameter >2 cm, clinically positive axillary lymph nodes not more than 2 (T2N1M0), Ki67≥+20%. Endocrine therapy sensitivity is defined as ER expression >50% by immunohistochemistry. HER-2 negativity is defined as HER-2 results of 0 or 1+ by immunohistochemistry, or negative by FISH;
3. Within 28 days before the first dose of study medication, patients must have at least one measurable lesion according to RECIST 1.1 standards, as assessed by ultrasound or MRI;
4. Laboratory test values: a. Absolute neutrophil count (ANC) ≥ 1,500/mm3 (1.5 × 10^9/L); b. Platelet count (PLT) ≥ 100,000/mm3 (100 × 10^9/L); c. Hemoglobin (Hb) ≥ 9 g/dL (90 g/L); d. Serum creatinine ≤ 1.5 times the upper limit of normal (ULN) or creatinine clearance ≥ 30 ml/min (based on the Cockroft-Gault formula); e. Total bilirubin (BIL) ≤ 1.5 times the upper limit of normal (ULN), Gilbert's syndrome; f. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) levels ≤ 2.5 times the upper limit of normal (ULN); g. INR or PT ≤1.5 ULN, APTT ≤1.5 ULN.
5. Subject agrees to collect tumor biopsy specimen during the screening period;
6. Subject signed the informed consent form, expressing willingness and ability to comply with the planned visits, study treatments, laboratory tests, and other trial procedures.

Exclusion Criteria:

1. Coexisted with other malignant tumors within 5 years prior to first medication, except for cured squamous cell carcinoma of the skin, basal cell carcinoma, non-muscle-invasive bladder cancer, carcinoma in situ of the cervix/breast, etc;
2. Had a serious infection within 1 month before screening or required systemic treatment for any active infection within 2 weeks before first medication;
3. History or current presence of autoimmune diseases, including but not limited to Crohn's disease, ulcerative colitis, systemic lupus erythematosus, sarcoidosis, Wegener's syndrome (granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis), autoimmune hepatitis, systemic sclerosis (scleroderma, etc.), Hashimoto's thyroiditis (exceptions are noted below), autoimmune vasculitis, autoimmune neuropathy (Guillain-Barre syndrome), etc. The following exceptions apply: Type I diabetes, thyroid dysfunction requiring only hormone replacement therapy (including thyroid dysfunction caused by autoimmune thyroid disease), psoriasis or vitiligo not requiring systemic treatment;
4. History of organ transplantation or allogeneic hematopoietic stem cell transplantation;
5. Patients who received systemic anti-cancer treatment within 2 weeks before the first dose, including chemotherapy, immunotherapy, hormone therapy, biological therapy (cytokines or growth factors that control the progression of cancer);
6. Metastatic breast cancer;
7. Positive for human immunodeficiency virus antibodies (HIV-Ab) or syphilis antibodies (Anti-TP); positive for hepatitis C virus antibodies (HCV-Ab), with hepatitis C virus RNA quantification > the upper limit of the normal value of the detection unit; positive for hepatitis B surface antigen (HBsAg) and/or hepatitis B core antibodies (HBcAb), with HBV DNA quantification > the lower limit of detection of the detection unit;
8. History of alcohol abuse or drug abuse.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
1. The proportion of (PEPI score 0 + pCR) in patients with discordant EPclin scores and Ki67 assessments who were randomly assigned to the "+CDK4/6i" group | Start of treatment until 6-month follow-up
  proportion of subjects who were PEPI score 0 or pCR after neoadjuvant endocrine therapy in patients with discordant EPclin scores and Ki67 assessments who were randomly assigned to the "+CDK4/6i" group

SECONDARY OUTCOMES:
The change in Ki-67 compared to the baseline after two weeks of treatment | Start of treatment until 2-week follow-up
The change in Ki-67 after surgery compared to two weeks post-treatment | Start of treatment until 6-month follow-up
Rate of patients with pCR (pathological complete response) after surgery | Start of treatment until 6-month follow-up
ORR | Start of treatment until 6-month follow-up
  Objective response rate: proportion of subjects who achieved complete remission (CR) or partial remission (PR) by primary tumor imaging evaluation
CCCA rate | Start of treatment until 6-month follow-up
  Cell cycle arrest: defined as Ki-67≤2.7%
Breast conservation rate | Start of treatment until 6-month follow-up
The proportion of PEPI 0-1 in patients with gene-high risk who are sensitive to single-agent AI treatment for two weeks and treated with AI in combination with Dalpiciclib | Start of treatment until 6-month follow-up
The proportion of PEPI 0-1 in patients with gene-low risk who are insensitive to single-agent AI treatment for two weeks and treated with AI in combination with Dalpiciclib | Start of treatment until 6-month follow-up
The proportion of patients at high risk according to Epclin who are downgraded to low risk after neoadjuvant treatment | Start of treatment until 6-month follow-up
EFS | Start of treatment until 24-month follow-up
  Event free survival: time from the start of treatment to the first occurrence of any of the following events: disease progression, local or distant recurrence, or death due to any cause
Incidence of adverse events (AE) | Start of treatment until 6-month follow-up
Incidence of serious adverse events (SAE) | Start of treatment until 6-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoqing Fan, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No